CLINICAL TRIAL: NCT00513357
Title: A Randomized Clinical Trial of Melatonin Versus Placebo and the Effect on Appetite in Advanced Cancer Patients
Brief Title: Melatonin Versus Placebo and the Effect on Appetite in Advanced Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2005-0901
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Results first posted 2012-09-14 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Gastrointestinal Cancer; Lung Cancer
Keywords: Gastrointestinal Cancer; Lung Cancer; Cachexia; Melatonin; Placebo; Anorexia; Weight Loss
MeSH Terms: conditions — Gastrointestinal Neoplasms; Lung Neoplasms; Cachexia; Anorexia; Weight Loss | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin (Experimental): 20 mg of Melatonin before going to sleep at night for a period of 4 weeks.
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): 20 mg of Placebo before going to sleep at night for a period of 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — 20 mg by mouth daily for 4 Weeks
  Arms: Melatonin
Drug: Placebo — Capsule by mouth daily for 4 Weeks
  Arms: Placebo

SUMMARY:
The goal of this clinical research study is to evaluate the effectiveness of melatonin for the management of poor appetite and weight loss in advanced cancer patients. The effectiveness of melatonin on weight gain, keeping/gaining of lean muscle mass, improved appetite, and side effects will also be evaluated.

DETAILED DESCRIPTION:
Melatonin is a hormone that is made by the part of the brain called the pineal gland and may help in letting your body know when it is time to go to sleep and when it is time to wake up. The researchers feel melatonin might help to improve your appetite, improve your overall sense of well-being, and maintain your current weight.

If you are found to be eligible to take part in this study, you will see a nutritionist at the first (baseline) visit. The nutritionist will measure the amount of calories you consume. You will be asked to report all food and drinks you have had in a 3-day period. If you are unable to remember what you have eaten and drunk in the last 3 days, you will be asked by the nutritionist to list all the food and drinks you have had within the last 24 hours.

Your arm muscle diameter and your skin fold below your shoulder blade will be measured on the arm you don't normally use to write with. This is to determine your body fat, lean mass and water content of your body.

Your resting energy expenditure will be measured. You will be asked to wear a breathing mask and to blow into a tube. This will allow your breath to be analyzed, to measure how many calories your body is using while you are at rest.

Blood (about 1-2 tablespoons) will be drawn for tests to make sure there are no other treatable causes for your weight loss.

This blood test may not need to be repeated if you have had a blood test in the last 3 months.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to one of 2 groups. Participants in Group 1 will take melatonin daily before bedtime for 4 weeks. Patients in Group 2 will take a placebo daily before bedtime for 4 weeks. A placebo is a substance that looks like the study drug but which has no active ingredients. You will have an equal chance (50/50) of being placed in either group. Neither you nor any of the medical staff or researchers on this study will know if you are receiving the study drug or placebo.

On Week 2, you will return to the clinic and you will repeat all the tests done at the baseline visit. If you are unable to return to M. D. Anderson to complete the evaluations on Day 14 (± 2 days), the research nurse will contact you by telephone and ask you about any side effects you are experiencing.

At Week 4, you will return to the clinic and all the tests done at baseline will be repeated.

At the end of 4 weeks, all study patients in both groups will be given the opportunity to take melatonin before going to sleep at night for an additional 4 weeks. If you choose not to continue on melatonin for an additional 4 weeks, you will be taken off study and blood will be drawn for your end of study tests which include albumin, C-reactive protein (CRP), thyroid stimulating hormone (TSH), vitamin B-12, and cortisol. These tests will require about 1-2 tablespoons of blood to be drawn. If you choose to continue on melatonin for an additional 4 weeks, you will be asked to return to the outpatient clinic at Week 6 to repeat the tests done at baseline.

Your end of study tests will be done at the end of 8 weeks.

You will continue to visit the study doctor at the outpatient clinic as long he feels it is necessary. At these visits, your height and weight will be recorded and you will be asked what food and drinks you have had.

This is an investigational study. Melatonin is not currently approved by the FDA except to treat blind people with no light perception for sleep disorders-and is considered a food/nutritional supplement. Up to 126 patients will be enrolled at MD Anderson and at Duke University Medical Center in Durham, North Carolina.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with solid gastrointestinal tumors or lung cancer patients referred to palliative care and a 5% or more involuntary weight loss within the last 6 months with anorexia (>3 on visual analog scale such as ESAS)
2. Greater than or equal to 18 years of age
3. Karnofsky score of 40 or higher
4. Patient has the ability to maintain oral food intake during the study period
5. If patients who have persistent anorexia/cachexia and are currently taking Megace, corticosteroids, non-steroidal anti-inflammatories (NSAID's), or thalidomide, they should be on the medication at least 2 weeks prior to study inclusion
6. Ability to sign informed consent and understand study procedures
7. Patient can continue all medications including complementary therapies or antineoplastic therapy while on-study other than melatonin if they have been on stable dose for at least 2 weeks
8. Negative pregnancy testing in women with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization.
9. Patients who cannot take Megace because of past history or elevated risk of DVT, adrenal insufficiency, impotence, hyperglycemia, CHF, menorrhagia, etc.
10. Patients who have persistent anorexia/cachexia after treatment with Megace has failed

Exclusion Criteria:

1. Patients who have dementia or delirium on entry into study as determined by the palliative care specialist using DSM-IV-criteria
2. Patients who are currently taking melatonin
3. Inability to take oral food during the study period
4. Unstable secondary cachexia caused by nausea, diarrhea, taste abnormalities, mucositis, constipation, dysphagia, or clinical depression prior to study inclusion. These symptoms should be resolved or stable for >/= 2 weeks at the time of inclusion into study as determined by the Palliative Care Specialist.
5. Inability to sign informed consent or understand study procedures
6. Karnofsky score of < 40
7. Patients < 18 years of age
8. Patients with </= 5% involuntary weight loss within the last 6 months and anorexia of < 3 on ESAS
9. Patients who are on complementary therapies containing melatonin or on medications for < 2 weeks and not on stable dose
10. Patients who have a cortisol level of </= 4.3 mg/dL at baseline will be excluded, unless they are on replacement corticosteroids.
11. Patients with a TSH of </= 0.50 or >/= 10 mcL/mL at baseline will be excluded
12. Pregnant females or females who are lactating/nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2006-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rony Dev, DO, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Joan Karnell Cancer Center, Philadelphia, Pennsylvania
  - UT MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Del Fabbro E, Dev R, Hui D, Palmer L, Bruera E. Effects of melatonin on appetite and other symptoms in patients with advanced cancer and cachexia: a double-blind placebo-controlled trial. J Clin Oncol. 2013 Apr 1;31(10):1271-6. doi: 10.1200/JCO.2012.43.6766. Epub 2013 Feb 25. PMID 23439759
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 07/21/2006 -04/08/2011. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Of the 125 participants, there were 52 participants excluded (43 did not meet inclusion criteria; and 9 declined to participate).
Period: Overall Study
Arm/Group | Melatonin | Placebo
Started | 38 | 35
Completed | 23 | 25
Not Completed | 15 | 10
Not completed — did not receive allocated placebo | 2 | 3
Not completed — Adverse Event | 4 | 2
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Disease Progression | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Melatonin | Placebo | Total
Number analyzed (Participants) | 38 | 35 | 73
Age Continuous [Mean (Full Range); unit: years]
  Age range | 59 [36 to 76] | 62 [32 to 86] | 59 [32 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 26 | 20 | 46
Region of Enrollment [Number; unit: participants]
  United States | 38 | 35 | 73

OUTCOME MEASURES:

1. Primary Outcome: Change in Appetite as Measured by ESAS
Description: Difference in ESAS (Edmonton Symptom Assessment Scale) assessment scores of appetite (symptom) from baseline evaluation [± 3 days] to 4 week evaluation [± 3 days], where the severity at the time of assessment is rated from 0 to 10 on a numerical scale; with 0 meaning that the symptom is absent and 10 that it is the worst possible severity.
Time Frame: Baseline and at 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 23 | 25
units on a scale | -0.83 (2.6) [6 to 8] | -1.19 (2.3) [4 to 9]

ADVERSE EVENTS:
Time Frame: 4 years and 2 months
Arm/Group | Melatonin | Placebo
Serious Adverse Events (participants affected / at risk) | 2/38 | 2/35
Other Adverse Events (participants affected / at risk) | 6/38 | 15/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melatonin (N=38) | Placebo (N=35)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 0 (0)
Alkaline Phosphatase (Investigations) | 0 (0) | 1 (1)
AST, SGOT (Investigations) | 0 (0) | 1 (1) — Aspartate transaminase (AST), serum glutamic oxaloacetic transaminase (SGOT)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Melatonin (N=38) | Placebo (N=35)
Confusion (Psychiatric disorders) | 1 (1) | 0/34 (0)
Fatigue (General disorders) | 1 (1) | 4/34 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 2/34 (2)
Pain (General disorders) | 0 (0) | 3/34 (3) — Abdomen
Somnolence (Nervous system disorders) | 1 (1) | 1/34 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0/34 (0)
Constitutional Symptom (other) (General disorders) | 0 (0) | 1/34 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1/34 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1/34 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1/34 (1)
Pain (General disorders) | 1 (1) | 0/34 (0)
Syncope (Fainting) (Nervous system disorders) | 0 (0) | 1/34 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes